CLINICAL TRIAL: NCT03616522
Title: A Prospective Study of Electronic Symptom Reporting Via Mobile Phone Among Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 03518
Record Dates: First submitted 2018-08-01; First posted 2018-08-06 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: a novel mobile phone-based intervention for automated electronic PRO collection — Over the three-month study period, patients will be prompted weekly via text message to self-report up to eleven common symptoms, as well as their performance status and quality of life.

SUMMARY:
Symptoms are common among patients with advanced malignancy undergoing treatment, and yet often go unrecognized by treatment providers. In addition to contributing to morbidity, poorly controlled symptoms drive emergency room utilization and hospital admission in this population, representing significant cost to patients, families, and the health care system. Systematic collection of patient-reported outcomes (PROs) has been proposed as a way to arm providers with the information necessary to intervene early, intensify symptom management, and improve symptom control. Recent research suggests that a standardized, web-based program of weekly patient-reported symptom monitoring leads to improved health-related quality of life and reduced acute care utilization; it may also prolong overall survival. Despite mounting evidence supporting its use among oncology patients, systematic PRO collection is lacking at most cancer centers, and optimal models for collection of PROs are poorly understood. The objective of this study is to evaluate prospectively the feasibility of a novel mobile phone-based intervention of weekly symptom reporting, among patients undergoing treatment for advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age ≥ 18 years) with advanced (metastatic) non-small cell lung cancer, initiating a new line of palliative-intent treatment at Abramson Cancer Center
* Ability to read and respond to questions in English
* Ability to provide informed consent to participate in the study
* Access to a smart phone capable of SMS-text messaging and internet access

Exclusion Criteria:

* Inability to read and respond to questions in English
* Inability or unwillingness to provide informed consent to participate in the study
* Inability to engage with SMS-text based platform
* Current enrollment in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced non-small cell lung cancer
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Number of subjects who will adhere to the mobile phone-based intervention | 3 months
  evaluate subjects to study-level adherence of a mobile phone-based intervention for automated PRO collection

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Shulman, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided